CLINICAL TRIAL: NCT00697203
Title: A Randomized, Double-blind Study of the Effect of RO4607381 in Combination With Pravastatin on HDL-cholesterol (HDL-C) Levels in Patients With Low or Average HDL-C Levels
Brief Title: A Study to Assess the Effect of RO4607381 in Patients With Relatively Low Levels of High Density Lipoprotein-Cholesterol (HDL-C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC18589
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Pravastatin; dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Dalcetrapib 300mg (Experimental)
  Interventions: Drug: Pravastatin; Drug: Dalcetrapib
- Dalcetrapib 600mg (Experimental)
  Interventions: Drug: Pravastatin; Drug: Dalcetrapib
- Dalcetrapib 900mg (Experimental)
  Interventions: Drug: Pravastatin; Drug: Dalcetrapib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Pravastatin

INTERVENTIONS:
Drug: Placebo — po daily for 12 weeks
  Arms: Placebo
Drug: Pravastatin — 40mg po daily for 12 weeks
Drug: Dalcetrapib — 300mg po daily for 12 weeks
  Arms: Dalcetrapib 300mg
Drug: Dalcetrapib — 600mg po daily for 12 weeks
  Arms: Dalcetrapib 600mg
Drug: Dalcetrapib — 900mg po daily for 12 weeks
  Arms: Dalcetrapib 900mg

SUMMARY:
This 4 arm study will evaluate the efficacy and safety of RO4607381 when co-administered with pravastatin in patients with low or relatively low HDL-C levels. Patients will be randomised to one of 4 groups to receive either RO4607381 300mg, 600mg or 900mg po daily, or placebo po daily, for 12 weeks.All patients will also receive pravastatin 40mg po daily for 12 weeks.The anticipated time on study treatment is 3 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-75 years of age;
* dyslipidemic patients with low or relatively low HDL-C levels during treatment with pravastatin.

Exclusion Criteria:

* women who are pregnant, breastfeeding, or of child-bearing potential;
* morbid obesity;
* uncontrolled hypertension;
* poorly controlled or insulin-treated diabetes;
* high creatinine levels or history of statin-associated myopathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (33):
  - Mobile, Alabama
  - Scottsdale, Arizona
  - Newark, Delaware
  - Miami, Florida
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Chalmette, Louisiana
  - Slidell, Louisiana
  - Auburn, Maine
  - Scarborough, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Towson, Maryland
  - St Louis, Missouri
  - Concord, New Hampshire
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Springdale, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Warminster, Pennsylvania
  - Fort Worth, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Started | 76 | 68 | 74 | 74
Completed | 67 | 62 | 66 | 67
Not Completed | 9 | 6 | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo | Total
Number analyzed (Participants) | 76 | 68 | 74 | 74 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.24) | 57.1 (10.53) | 56.7 (10.52) | 57.2 (10.87) | 56.7 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 17 | 15 | 58
  Male | 63 | 55 | 57 | 59 | 234

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in HDL-C Level\n
Time Frame: Week 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Number analyzed (Participants) | 75 | 67 | 72 | 73
mg/dL | 17.18 (2.19) | 31.42 (2.29) | 36.45 (2.24) | 2.31 (2.18)

2. Primary Outcome: Percent Change From Baseline in HDL-C Level\n
Time Frame: 12 Weeks
Measure: Least Squares Mean (Standard Error); unit: Percent change in mg/dL
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Number analyzed (Participants) | 75 | 67 | 72 | 73
Percent change in mg/dL | 6.58 (0.84) | 11.90 (0.88) | 13.92 (0.86) | 0.73 (0.84)

3. Secondary Outcome: Change From Baseline in: Total Cholesterol, Triglycerides, HDL-C, LDL-C, HDL-2, HDL-3, ApoA1, ApoA2, ApoB, LpAI
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Percent change in mg/dL
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Number analyzed (Participants) | 76 | 68 | 74 | 74
Percent change in mg/dL
  Total Cholesterol | 7.08 (1.45) | 12.58 (1.52) | 9.36 (1.48) | 1.35 (1.45)
  Triglycerides | -5.95 (3.93) | 4.45 (4.11) | -5.01 (4.02) | -4.25 (3.93)
  HDL-C | 17.18 (2.19) | 31.42 (2.29) | 36.45 (2.24) | 2.31 (2.18)
  LDL-C | 8.51 (2.58) | 10.88 (2.73) | 5.28 (2.65) | 3.84 (2.59)
  HDL-2 | 52.10 (8.19) | 97.40 (8.82) | 121.2 (8.49) | 10.54 (8.86)
  HDL-3 | 11.95 (1.96) | 20.94 (2.11) | 23.56 (2.03) | 0.68 (2.12)
  ApoA1 | 7.03 (1.39) | 13.60 (1.44) | 14.90 (1.40) | 1.01 (1.46)
  ApoA2 | 3.82 (1.23) | 8.07 (1.33) | 8.36 (1.28) | 0.72 (1.33)
  ApoB | 2.66 (1.90) | 4.62 (2.01) | -1.64 (1.95) | -0.71 (1.98)
  LpA1 | 15.06 (3.59) | 22.68 (3.59) | 24.76 (3.40) | 3.32 (3.81)

4. Secondary Outcome: Percent Change of Fasting Glucose Level
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Percent change in mg/dL
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Number analyzed (Participants) | 76 | 68 | 74 | 74
Percent change in mg/dL | 3.61 (1.69) | 6.03 (1.79) | 5.42 (1.72) | 3.00 (1.70)

5. Secondary Outcome: AEs, Lab Parameters, Vital Signs, ECG
Time Frame: Through 9 Months
Population: Data not collected
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Ratios of Total HDL-C/LDL-C, HDL-2/HDL-3, ApoA1/ApoB
Time Frame: Baseline and at 12 Weeks
Measure: Least Squares Mean (Standard Error); unit: Percent Change in Ratio
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Number analyzed (Participants) | 75 | 67 | 72 | 73
Percent Change in Ratio
  HDL-C/LDL-C | -3.76 (2.96) | -16.0 (3.20) | -19.4 (3.04) | 3.09 (2.95)
  ApoB/ApoA1 | -4.97 (2.10) | -5.79 (2.19) | -12.7 (2.11) | -1.84 (2.50)
  HDL-2/HDL-3 | 35.18 (5.88) | 63.40 (6.33) | 76.38 (6.10) | 8.89 (6.37)

ADVERSE EVENTS:
Arm/Group | Dalcetrapib 300mg | Dalcetrapib 600mg | Dalcetrapib 900mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/76 | 2/68 | 3/74 | 2/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/68 | 0/74 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib 300mg (N=76) | Dalcetrapib 600mg (N=68) | Dalcetrapib 900mg (N=74) | Placebo (N=74)
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No